CLINICAL TRIAL: NCT04002284
Title: The Efficacy and Safety of Anlotinib in Metastatic HER2 Negative Breast Cancer, a Single Arm Phase II Clinical Trial
Brief Title: Anlotinib in Metastatic HER2 Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peng Yuan (Unknown)
Responsible Party: Sponsor-Investigator, Peng Yuan, chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC1692
Record Dates: First submitted 2019-06-23; First posted 2019-06-28 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Breast Neoplasm; Antineoplastic Agents; Anlotinib
MeSH Terms: conditions — Breast Neoplasms | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anlotinib (Experimental): anlotinib 12mg qd p.o. d1-14/21day/cycle
  Interventions: Drug: Anlotinib Hydrochloride

INTERVENTIONS:
Drug: Anlotinib Hydrochloride — Anlotinib 12mg p.o. d1-14, 21days/cycle
  Other Names: anlotinib

SUMMARY:
The hypothesis of this study is to discover if the anlotinib can shrink or slow the growth of pretreated HER2 negative metastatic breast cancer.

DETAILED DESCRIPTION:
Breast cancer is one of the most common malignant tumors in women, which is a serious threat to women's health. Despite the continuous improvement of treatment, 30% of breast cancer eventually develops into advanced breast cancer. The median survival of advanced breast cancer after routine treatment is 2-3 years. The main treatments include chemotherapy, endocrine therapy, and targeted therapy. The treatment of metastatic breast cancer (MBC) aims to improve quality of life, reduce pain and prolong survival.

Angiogenesis plays an important role in tumor cell proliferation and metastasis. Various anti-angiogenic drugs such as bevacizumab, sunitinib, sorafenib, etc. have been developed and widely used in various tumors. Treatments such as colon cancer, lung cancer, and renal cell carcinoma significantly improve PFS and OS in patients with advanced disease, and the adverse reactions are well tolerated. However, anti-angiogenic therapy has certain limitations in the treatment of advanced breast cancer.

Anrotinib hydrochloride capsule is a new drug independently developed in China. It is a multi-target receptor tyrosine kinase inhibitor targeting angiogenesis-related kinases such as VEGFR1/2/3, FGFR1/2/3 and other kinases such as cell growth-related kinases such as PDGFRα/β, c-Kit, and Ret , and it was approved by China Food and Drug Administation for the treatment of patients with locally advanced or metastatic non-small cell lung cancer who have progressed or relapsed after receiving at least 2 systemic chemotherapy. Basic research shows that anlotinib is effective in breast cancer cell lines, but lacks the results of clinical application of advanced breast cancer. This study is based on the results of phase I clinical trials of allerinib in a variety of advanced solid tumors, to explore its efficacy and safety in HER2-negative advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 year-old women; Pathologically or cytologically confirmed breast cancer; HER2 negative(immunohistochemistry or fluorescence in situ hybridization);
* ECOG score: 0-1, expected survival time ≥ 3months;
* Anthracycline- / taxane- pretreated (adjuvant, neoadjuvant) breast cancer patients who have failed from 1-2 standard chemotherapies after recurrence and metastasis;
* According to RECIST 1.1, exist at least ≥1 measurable lesion(CT >1cm，other examination >2cm);
* The patients have enough organ function. The laboratory test indexes must comply with the following requirements:

Blood routine: neutrophil≥1.5G/L, platelet count ≥80G/L, hemoglobin ≥90g/L Liver function: serum bilirubin ≤ 1.5 times the upper limit of normal value; ALT and AST≤2.5 times the upper limit of normal value; ALT and AST≤5 times the upper limit of normal value when liver metastasis Renal function: serum creatinine ≤ 1.0times the upper limit of normal value, creatinine clearance >50ml/min（Cockcroft-Gault formula)

* Women of child-bearing age should be carried out pregnancy test (serum or urine) within 7 days before recruit, the results should be negative; and are willing to adopt the appropriate methods of contraception during the trial and 8 weeks after last administration；
* Can swallow oral drugs;
* The patients have good compliance to the therapy and follow-up to be scheduled and are able to understand the study protocol and sign the Informed Consent Form.

Exclusion Criteria:

* The patients in pregnancy or lactation growth period and did not take effective contraception;
* The patients who received ≥3 chemotherapies（Do not include endocrine therapy）after recurrence and metastasis; involved in other clinical trials four weeks prior to the start of the study;
* The patients with a variety of factors that affect the oral administration and absorption of drugs;
* The patients with rapid progression of viscera invasion(liver lesion >1/2 viscera area or liver dysfunction);
* The patients have uncontrollable mental illness.
* The patients who had serious adverse effect to oral etoposide or were allergic to etoposide.
* The patients who have only bone metastasis without other measurable lesion;
* The patients experience severe cardiovascular diseases;
* The patients experience severe upper gastrointestinal ulcer or malabsorption syndrome.
* Abnormal bone marrow functions(neutrophil<1.5G/L, platelet count <75G/L, hemoglobin <90g/L);
* Abnormal renal function(serum creatinine > 1.5 times the upper limit of normal value);
* Abnormal liver function(serum bilirubin ≤ 1.5 times the upper limit of normal value);
* The patients have uncontrollable brain metastasis;
* The patients do not have good compliance to the therapy.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
objective response rate(ORR) | through study completion, an average of 1 year
  Objective response rate defined as confirmed complete response or partial response under RECIST 1.1 criteria. CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. To be assigned a status of CR or PR, changes in tumor measurements must be confirmed by repeat assessments performed no fewer than 4 weeks after the response criteria are first met.

SECONDARY OUTCOMES:
disease control rate(DCR) | through study completion, an average of 1 year
  Number of participants with stable disease or partial response or complete response treating by anloitnib according to RESIST criteria v1.1.
Progression free survival (PFS) | From date of enrollment until the date of first documented progression, assessed up to 24 months
  Progression-free survival estimated using Kaplan-Meier methods is defined as the time from the date of informed consent to the earlier of death or disease progression. Patients alive without disease progression are censored at the date of last disease evaluation. Progressive disease (PD) based on RECIST 1.1 is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Equivocal progression of non-target lesions also qualifies as PD.
overall survival(OS) | From date of enrollment until death, assessed up to 24 months
  OS, defined as the time from the date of informed consent until to the date of death, regardless of the cause of death.
Safety and Tolerability | through study completion, an average of 1 year
  All the treatment-related adverse events occurred as assessed by CTCAE v4.0

OTHER OUTCOMES:
circulating tumor DNA biomarker | From date of enrollment until the date of first documented progression, assessed up to 24 months
  biomarkers measurement in dynamic circulating tumor DNA sequencing on the day of enrollment and at the end of every two cycle (28 days one cycle)

CONTACTS AND LOCATIONS:
Overall Officials: Peng Yuan, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- National Cacner Center/ Cancer Hospital,Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No